CLINICAL TRIAL: NCT05504135
Title: Implementation of Pre-emptive Pharmacogenomics Testing in Singapore-based Private Hospital Institutions (IMPT Study)
Status: Completed | Type: Observational
Sponsor: Nalagenetics Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: SG-RMG-01-20190401
Record Dates: First submitted 2022-08-11; First posted 2022-08-17 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pre-emptive Pharmacogenomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- RMG Patients
  Interventions: Diagnostic Test: Pharmacogenomics Testing

INTERVENTIONS:
Diagnostic Test: Pharmacogenomics Testing — To test if pharmacogenomics information (produced from testing) included by us in the Raffles' Electronic Health Records (EHR) will be used by physicians to personalize patients' prescriptions.

SUMMARY:
In collaboration with Raffles Medical Group, we will be recruiting 500 patients and following them for the next 3-12 months to see whether pharmacogenomics information provided in the Raffles' Electronic Health Records (EHR) will be used by physicians to personalize patients' prescriptions.

DETAILED DESCRIPTION:
Pre-emptive genotyping provides relevant genomic data to physicians to facilitate prescribing and to facilitate checking of prescriptions by pharmacists to ensure drug safety and efficacy. This essential information should be incorporated into electronic healthcare systems and should be readily available. The effectiveness of pre-emptive genotyping to reduce adverse drug reactions (ADRs) is unknown in Singapore. Hence, this study is designed to evaluate whether it is feasible to implement large scale pre-emptive genotyping program at a hospital in Singapore and aim to integrate genomic medicine into clinical practice to improve drug safety and efficacy.

This study involves the testing of feasibility of pharmacogenomic genotyping in hospitals whereby our pharmacogenomics panel tests for 5 genes (CYP2D6, CYP2C9, CYP2C19, SLCO1B1 and HLA-B*58:01) which influences patient's response to more than 165 medications. Reports will be generated for all drugs that have been reported to be in CPIC Level A/B of association with the genes/haplotypes. The patients who are given these tests for free are recommended due to having experienced at least one of the diseases in our list or is at a risk of developing them.

ELIGIBILITY:
Inclusion Criteria:

* Patients who experienced at least one of the following diseases, or is at risk of developing them:

  1. Diabetes Mellitus
  2. Hypertension
  3. Hyperlipidaemia
  4. Ischaemic Heart Disease
  5. Stroke
  6. Osteoarthritis
  7. Rheumatoid Arthritis
  8. Gout
  9. Anxiety
  10. Major Depression

      Exclusion Criteria:
* Below ages 21 and above ages 65

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250 patients visiting Raffles Hospital in Singapore
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Turnaround time of genotype result, compared to expected | 6 months
Overall satisfaction of patient | 0 months
  Via survey upon recruitment
Overall satisfaction of patient | 3 month
  Via survey at month 3 of the study
Overall satisfaction of patient | 12 months
  Via survey at month 12 of the study
Overall satisfaction of site principal investigators | 6 months
  Via survey done at month 6 of the study
Overall satisfaction of prescribing physicians | 12 months
  Via survey done at month 12 of the study
Prevalence of clinically actionable genotypes | 12 months
  The number of patients receiving recommendations that includes a certain follow up action which includes monitoring, change of dosing or change of prescription.
Recommendation acceptance rate | 12 months
  Defined by: (1) Number of physicians who are interested to consider pharmacogenomics information to guide prescription, measured by click-through rate of Pharmacogenomics Access Button; (2) Number of changes made to the medications post-PGx testing; (3) Data obtained from satisfaction survey for prescribing physicians

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Wong, Dr, Principal Investigator — Raffles Medical Group
Locations (1):
- Raffles Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng FF, Verma R, Sani L, Irwanto A, Lee M, Wee A, Chng SK, Wong M, Chan A. A feasibility study on implementing pre-emptive pharmacogenomics testing in outpatient clinics in Singapore (IMPT study). Pharmacogenomics J. 2025 Mar 12;25(1-2):7. doi: 10.1038/s41397-025-00366-1. PMID 40074758